CLINICAL TRIAL: NCT04081402
Title: A Phase 1/3 Clinical Trial to Evaluate the Safety and Efficacy of HUTOX Compared to Botox® in Subjects With Moderate to Severe Crow's Feet Lines
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HU-014_P1/3_CFL
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Crow's Feet Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HU-014 Inj (Experimental)
  Interventions: Biological: HU-014
- Botox Inj (Active Comparator)
  Interventions: Biological: Botox Inj

INTERVENTIONS:
Biological: HU-014 — Hutox Inj(Clostridium botulinum type A)
  Arms: HU-014 Inj
Biological: Botox Inj — Botox Inj(Clostridium botulinum type A)
  Arms: Botox Inj

SUMMARY:
A Phase 1/3 Clinical Trial to Evaluate the Safety and Efficacy of HUTOX Compared to Botox® in Subjects With Moderate to Severe Crow's Feet Lines

ELIGIBILITY:
Inclusion Criteria:

* Bilaterally symmetrical moderate-to-severe CFL at maximum smile on the FWS as rated by the investigator

Exclusion Criteria:

* Volunteer who has history of any diseases following. (myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis etc.)
* From screening, Subject who get a plastic Surgery within 48 Weeks
* Subject who has skin disorder including infection and scar on injection site
* Subject who takes a medication including skeletal muscle relaxants, Aminoglycoside, lincomycin, anticholinergic drug, benzodiazepine, benzamide etc.
* Subject who takes a medication including anticoagulant, antithrombotic drug except low dose aspirin (below 325 mg/day)
* Any condition that, in the view of the investigator, would interfere with study participation

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of Crow's feet Lines improvement rate [Time Frame: Week 4] | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No